CLINICAL TRIAL: NCT02196142
Title: Acute Effects of Cortisol on Alcohol Craving in Alcohol Dependence
Acronym: CAR-Bern 2013
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 068/14
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Alcohol Craving; Psychological Stress; Physiological Stress
Keywords: Cortisol; Alcohol Craving; Alcohol Dependence
MeSH Terms: conditions — Stress, Psychological; Alcoholism | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cortisol first, Placebo second (Active Comparator): Drug: Cortisol 20mg, Drug: Mannitol (used as placebo)
  Interventions: Drug: Cortisol 20mg; Drug: Placebo Mannitol
- Placebo first, Cortisol second (Active Comparator): Drug: Cortisol 20mg, Drug: Mannitol (used as placebo)
  Interventions: Drug: Cortisol 20mg; Drug: Placebo Mannitol

INTERVENTIONS:
Drug: Cortisol 20mg — Drug: Cortisol 20mg
Drug: Placebo Mannitol — Drug: Placebo Mannitol

SUMMARY:
To investigate the effects of cortisol on alcohol craving and stress reactivity in alcohol addicted subjects.

Randomized, double-blind, placebo-controlled, cross-over, single administration of study medication.

Study hypothesis: Cortisol has an inhibiting effect on alcohol craving and stress reactivity in alcohol dependent subjects.

DETAILED DESCRIPTION:
Background

Alcohol dependence is a chronically and relapsing disorder with major impact on the persons psychological, physiological and social functioning. There is extensive evidence from animal and human studies pointing out the important role of addiction memory in the development and maintenance of the disorder.

Cognitive behavioural therapy (CBT) has proven its high effectiveness in the treatment for addictive disorders. A core element of CBT are exposure techniques that are comparable to extinction and habituation learning. The repeated exposure to alcohol related cues in the absence of alcohol ingestion will lead to extinction of conditioned responses, thus reducing the probability of relapse to alcohol taking behaviour.

Studies have shown that glucocorticoids impair memory retrieval in healthy subjects. In fact, the investigators could show that cortisol has a fear reducing effect in patients with post-traumatic stress disorder and in phobic patients, resulting particularly in reduced symptoms of anxiety and in reduced stress reactivity. Interestingly enough, pharmacologically induced high levels of glucocorticoids lowered the subjective feeling of anxiety and stress in situations activating per se the HPA-axis. Further it has been shown that the combined therapy of glucocorticoid administration and exposition based psychotherapy leads to better therapy outcome in patients with specific phobias.

Objective

The goal of this study is to examine the acute effects of glucocorticoids administration on alcohol craving and stress reactivity of abstinent alcohol dependent patients. On the basis of clinical research in anxiety disorders, the investigators expect that a pharmacologically increased cortisol level may impair the retrieval of addiction memory, which is indicated by less craving during the alcohol exposition, while exposition therapy enhances consolidation of corrective experiences. Similar to the research in anxiety patients, the investigators aim to examine whether cortisol administration could help improve the effects of exposition therapy in patients with alcohol dependence. The purpose is to decrease therapy duration through cortisol administration in addition to already well proven therapies and make the therapy more efficient as well as a factor in reducing healthcare costs.

Methods

Patients undergo two identical experimental sessions between the 6th and 8th week (one week in between) of their 12-week inpatient treatment program for alcohol dependence. The experiment takes place in the experimental rooms of the clinic Südhang between 1 and 6 pm. One hour before the confrontation with alcohol associated stimuli patients receive either 20mg of hydrocortisone or placebo (oral administration). The experiment consists of a computer based picture task (alcoholic and neutral pictures) and an in-vivo exposure task. Psychological (craving, stress, arousal) and physiological (heart rate, saliva cortisol) parameters are repeatedly measured over the course of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Abstinent alcoholics in the 12-week in-patient program of the Clinic Südhang
* Abstained from alcohol for at least 6 weeks
* Voluntarily signed informed consent

Exclusion Criteria

* Co-morbid psychiatric disturbances (such as major depression, bipolar disorder, schizophrenia)
* Current medical conditions excluding participation (such as acute infectious disease)
* Recent history of systemic or topic glucocorticoid therapy
* Known hypersensitivity to the IMP under investigation (cortisol)
* Pregnancy, breast-feeding
* Inability to read and understand the participant's information
* Positive alcohol test according to breathalyser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in alcohol craving score | During and after presentation of drug stimuli, expected to be after 10 minutes
  Measured by Alcohol Urge Questionnaire & Visual Analogue Scale

SECONDARY OUTCOMES:
Change from baseline in State-Trait-Anger Expression Inventory STAXI | After presentation of drug stimuli, expected to be after 20 minutes
Change from baseline in heart rate variability | During and after presentation of drug stimuli, expected to be after 10 minutes
Saliva Cortisol Level | After presentation of drug stimuli, expected to be after 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Leila Soravia, Dr. phil., Study Director — University Hospital of Psychiatry Bern; Peter Allemann, Dr. med., Principal Investigator — Clinic Südhang; Dominique de Quervain, Prof. Dr., Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- Klinik Südhang, Kirchlindach, Canton of Bern, Switzerland